CLINICAL TRIAL: NCT04816747
Title: Intradiscal and Intra-articular Injection of Autologous Platelet-Rich-Plasma (PRP) in Patients With Lumbar Degenerative Disc Disease and Facet Joint Syndrome: A Prospective, Single-arm, Open Label Clinical Trial
Brief Title: Intradiscal and Intra-articular Injection of Autologous Platelet-Rich-Plasma (PRP) in Patients With Lumbar Degenerative Disc Disease and Facet Joint Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Stylianos Kapetanakis (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor-Investigator, Stylianos Kapetanakis, Director of Spine Department and Deformities (Interbalkan European Medical Center, Thessaloniki, Greece) and Department of Minimally Invasive and Endoscopic Spine Surgery (Athens Medical Center, Athens, Greece), European Interbalkan Medical Center
Organization: European Interbalkan Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Not administered
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Degenerative Disc Disease; Facet Joint Syndrome
Keywords: Platelet-rich-plasma; intradiscal; intra-articular; degenerative disc disease; facet joint syndrome; facet joint arthritis
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: All participants fulfilling the predetermined inclusion criteria will be considered eligible to be subjected to treatment with PRP. Injection of PRP will be conducted intradiscally and/or intra-articularly, in cases of lumbar DDD and/or FJS, as defined by clinical and radiologic assessment. Hence, all participants will be assigned to the same intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous PRP (Experimental): Participants with diagnosed lumbar DDD are planned to be managed via intradiscal injection of 0.5-1 ml autologous PRP, whereas participants with FJS will be injected with 0.5 ml of respective solution. All procedures will be performed in surgical theatre under constant fluoroscopic guidance.
  Interventions: Biological: Autologous PRP

INTERVENTIONS:
Biological: Autologous PRP — Participants enrolled in this study will be managed with intradiscal and/or intra-articular injections of autologous PRP according to features of underlying pathology. Participants featuring FJS will be prior to PRP diagnostically and therapeutically injected with local anesthetic in order to verify FJS as the etiology of experienced pain. Injected PRP solution volume is designed to be 0.5-1 ml and 0.5 ml in cases of intradiscal and intra-articular injection, respectively. All participants are planned to receive a single dose of PRP, whilst a maximum of two compromised discs and four facet joints will be treated in each patient.

SUMMARY:
Autologous Platelet-Rich-Plasma (PRP) represents a regenerative therapy that has gained remarkable ground in the field of orthopaedics in recent years. PRP has been implemented for a plethora of musculoskeletal ailments, being associated with minor complications and noteworthy efficacy (Akeda et al., 2019). PRP has been depicted to contain a variety of growth factors crucial for regulation of cell proliferation and migration as well as extracellular matrix synthesis (Cheng et al., 2019). Furthermore, therapeutic effect of PRP administration is considered to be additionally exerted via its anti-inflammatory and immunoregulative properties, as it has been delineated to induce regional decrease of pro-inflammatory mediators at the injection site (Hirase et al., 2020).

Lumbar Degenerative Disc Disease (DDD) and Facet Joint Syndrome (FJS) constitute chronic degenerative conditions of lumbar spine that have been associated with substantial morbidity and disability in recent years. Besides the noted progress in comprehension of these conditions' pathogenesis, available therapeutic modalities remain extremely limited and controversial, being not capable of altering the natural progress of underlying disease (Wu et al., 2016; Wu et al., 2017; Hirase et al., 2020).

Autologous PRR has been recommended as a beneficial alternative instead of conventional treatment strategies for interventional management of lumbar DDD and FJS (Aufiero et al., 2015; Navani and Hames, 2015; Kirchner and Anitua, 2016; Levi et al., 2016; Tuakli-Wosornu et al., 2016; Wu et al., 2016; Akeda et al., 2017; Lutz GE, 2017; Wu et al., 2017; Cheng et al., 2019). Results of these studies indicated that intra-discal and intra-articular injection of PRP for DDD and FJS respectively is characterized by safety and satisfactory efficacy in reducing intensity of clinical manifestations, exerting also potentially regenerative effects. However, quality of available evidence is remarkably low, since in the overwhelming majority of these studies was a limited number of patients evaluated. Furthermore, determined follow-up intervals were not extended and, most importantly, patients were not majorly with rigorous clinical and radiologic criteria selected.

Aim of this study is to investigate the precise effects of intradiscal and intra-articular injection of PRP in patients with early-stage lumbar DDD and FJS, as determined by particular radiologic classifications. The prospective design, the defined greater number of recruited individuals in pilot analysis as well as the comparatively greater follow-up underline the originality of our protocol.

ELIGIBILITY:
Eligibility criteria will be distinctly applied in participants with lumbar DDD and FJS prior to treatment application.

A. Participants with lumbar DDD

Inclusion Criteria

* Recurring low back pain persistent for more than 6 months demonstrating discogenic origin (i.e. localized at midline, exacerbated in seated position and alleviated in bed rest)
* Failure of initially implemented conservative measures (medication regimen and/or physical therapy sessions or other injections)
* Imaginary findings of Grade I-III DDD according to radiologic MRI-based classification proposed by Pfirrmann et al. (Pfirrmann et al., 2001)
* Absence of exclusion criteria, as defined below.

Exclusion Criteria

* Presence of local or systemic infection signs (clinical and laboratory)
* Concurrent known systemic inflammatory disease with musculoskeletal manifestations or other chronic inflammatory disease
* Concurrent known hemorrhagic disorder or antithrombotic regimen
* Presence of Grade IV-V DDD according to Pfirrmann classification (Pfirrmann et al., 2001)
* Spondylolysis/Spondylolisthesis
* Intervertebral Disc Herniation
* Previous spinal surgery
* Spinal Stenosis
* Primary or Secondary spinal tumour
* Spinal fracture in past 6 months
* Diagnosed psychiatric disorder
* Epidural steroid or other intradiscal injection or within past 30 days
* Administration of NSAIDs, steroids or dietary supplements with anti-inflammatory properties within past 30 days.

Β. Participants with lumbar FJS

Inclusion Criteria

* Recurring low back pain persistent for more than 6 months with no radiation to buttock or lower limb, presence of exacerbation in lateral bending, rotation and extension and paraspinal localization featuring reproduction with pressure.
* Failure of conservative treatment measures (medication regimen and/or physical therapy sessions or other injections).
* Radiologic findings of Grade I-II FJS according to CT-based classification proposed by Suri et al. (Suri et al., 2010)
* Absence of exclusion criteria, as designated below.

Exclusion Criteria

* Clinical manifestations of radiculopathy
* Presence of local or systemic infection signs (clinical and laboratory)
* Concurrent known systemic inflammatory disease with musculoskeletal manifestations or other chronic inflammatory disease
* Concurrent known hemorrhagic disorder or antithrombotic regimen.
* Presence of Grade III-IV FJS according to proposed classification of Suri et al. (Suri et al., 2010)
* Spondylolysis/Spondylolisthesis
* Intervertebral Disc Herniation
* Previous spinal surgery
* Spinal Stenosis
* Primary or Secondary spinal tumour
* Spinal fracture in past 6 months
* Diagnosed psychiatric disorder
* Previous intra-articular steroid injection within past 30 days
* Administration of NSAIDs, steroids or dietary supplements with anti-inflammatory properties within past 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain Visual Analogue Scale (VAS) Scores from baseline to post intervention during follow-up | VAS score is planned to be evaluated preoperatively, immediately after intervention, at 6 weeks and at 3,6,12 and 24 months postoperatively.
  Participants will be asked to indicate the pain level according to their subjective perception with as spot in a unipolar horizontal line of 100 mm (0: no pain, 100: the worst pain possible). Scores will be calculated in mm, and an one-decimal place approach will be adopted for record.
Alteration in Short-Form 36 (SF-36) Medical Health Survey Questionnaire Scores from baseline to post intervention during follow-up | SF-36 questionnaire is planned to be evaluated preoperatively, immediately after intervention, at 6 weeks and at 3,6,12 and 24 months postoperatively.
  Participants will be asked to complete the analogous questionnaire, so that eight distinct parameters reflecting general health status are evaluated: physical function (PF), role-physical (RP), bodily pain (BP), general health (GH), energy, fatigue and vitality (V), social function (SF), role-emotional (RE) and mental health (MH). Computational processing of collected data will be subsequently conducted, so that each parameter is expressed by a percentage. Greater scores in these 8 parameters are associated with ameliorated Health-Related Quality of Life (HRQoL).

SECONDARY OUTCOMES:
Complications | Complications will be constantly recorded during the study immediately after intervention, at 6 weeks and at 3,6,12 and 24 months postoperatively.
  Safety of implemented procedure is designed to be determined via the record of frequency and kind of perioperative associated complications.

CONTACTS AND LOCATIONS:
Overall Officials: Stylianos Kapetanakis, Assistant Professor, Principal Investigator — Spine Department and Deformities, Interbalkan European Medical Center, Thessaloniki, PC 55535, Greece; Department of Minimally Invasive and Endoscopic Spine Surgery, Athens Medical Center, Athens, PC 15124, Greece; Nikolaos Gkantsinikoudis, PhD Candidate, Study Chair — Spine Department and Deformities, Interbalkan European Medical Center, Thessaloniki, PC 55535, Greece; Aristeidis Kritis, Associate Professor, Study Chair — Department of Physiology and Pharmacology, School of Medicine, Faculty of Health Sciences, Aristotle University of Thessaloniki (A.U.Th), Thessaloniki, PC 54124, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akeda K, Yamada J, Linn ET, Sudo A, Masuda K. Platelet-rich plasma in the management of chronic low back pain: a critical review. J Pain Res. 2019 Feb 25;12:753-767. doi: 10.2147/JPR.S153085. eCollection 2019. PMID 30881089
- [Background] Cheng J, Santiago KA, Nguyen JT, Solomon JL, Lutz GE. Treatment of symptomatic degenerative intervertebral discs with autologous platelet-rich plasma: follow-up at 5-9 years. Regen Med. 2019 Sep;14(9):831-840. doi: 10.2217/rme-2019-0040. Epub 2019 Aug 29. PMID 31464577
- [Background] Hirase T, Jack Ii RA, Sochacki KR, Harris JD, Weiner BK. Systemic Review: Is an Intradiscal Injection of Platelet-Rich Plasma for Lumbar Disc Degeneration Effective? Cureus. 2020 Jun 25;12(6):e8831. doi: 10.7759/cureus.8831. PMID 32607308
- [Background] Wu J, Du Z, Lv Y, Zhang J, Xiong W, Wang R, Liu R, Zhang G, Liu Q. A New Technique for the Treatment of Lumbar Facet Joint Syndrome Using Intra-articular Injection with Autologous Platelet Rich Plasma. Pain Physician. 2016 Nov-Dec;19(8):617-625. PMID 27906940
- [Background] Wu J, Zhou J, Liu C, Zhang J, Xiong W, Lv Y, Liu R, Wang R, Du Z, Zhang G, Liu Q. A Prospective Study Comparing Platelet-Rich Plasma and Local Anesthetic (LA)/Corticosteroid in Intra-Articular Injection for the Treatment of Lumbar Facet Joint Syndrome. Pain Pract. 2017 Sep;17(7):914-924. doi: 10.1111/papr.12544. Epub 2017 Feb 22. PMID 27989008
- [Background] Aufiero D, Vincent H, Sampson S, Bodor M. Regenerative Injection Treatment in the Spine: Review and Case Series with Platelet Rich Plasma. J Stem Cells Res, Rev & Rep. 2015;2(1):1019.
- [Background] Levi D, Horn S, Tyszko S, Levin J, Hecht-Leavitt C, Walko E. Intradiscal Platelet-Rich Plasma Injection for Chronic Discogenic Low Back Pain: Preliminary Results from a Prospective Trial. Pain Med. 2016 Jun;17(6):1010-22. doi: 10.1093/pm/pnv053. Epub 2015 Dec 26. PMID 26814283
- [Background] Kirchner F, Anitua E. Intradiscal and intra-articular facet infiltrations with plasma rich in growth factors reduce pain in patients with chronic low back pain. J Craniovertebr Junction Spine. 2016 Oct-Dec;7(4):250-256. doi: 10.4103/0974-8237.193260. PMID 27891035
- [Background] Navani A, Hames A. Platelet-rich plasma injections for lumbar discogenic pain: A preliminary assessment of structural and functional changes. Techniques in Regional Anesthesia and Pain Management 2015;19(1-2):38-44.
- [Background] Tuakli-Wosornu YA, Terry A, Boachie-Adjei K, Harrison JR, Gribbin CK, LaSalle EE, Nguyen JT, Solomon JL, Lutz GE. Lumbar Intradiskal Platelet-Rich Plasma (PRP) Injections: A Prospective, Double-Blind, Randomized Controlled Study. PM R. 2016 Jan;8(1):1-10; quiz 10. doi: 10.1016/j.pmrj.2015.08.010. Epub 2015 Aug 24. PMID 26314234
- [Background] Akeda K, Ohishi K, Masuda K, Bae WC, Takegami N, Yamada J, Nakamura T, Sakakibara T, Kasai Y, Sudo A. Intradiscal Injection of Autologous Platelet-Rich Plasma Releasate to Treat Discogenic Low Back Pain: A Preliminary Clinical Trial. Asian Spine J. 2017 Jun;11(3):380-389. doi: 10.4184/asj.2017.11.3.380. Epub 2017 Jun 15. PMID 28670405
- [Background] Lutz GE. Increased Nuclear T2 Signal Intensity and Improved Function and Pain in a Patient One Year After an Intradiscal Platelet-Rich Plasma Injection. Pain Med. 2017 Jun 1;18(6):1197-1199. doi: 10.1093/pm/pnw299. No abstract available. PMID 28339718
- [Background] Pfirrmann CW, Metzdorf A, Zanetti M, Hodler J, Boos N. Magnetic resonance classification of lumbar intervertebral disc degeneration. Spine (Phila Pa 1976). 2001 Sep 1;26(17):1873-8. doi: 10.1097/00007632-200109010-00011. PMID 11568697
- [Background] Suri P, Katz JN, Rainville J, Kalichman L, Guermazi A, Hunter DJ. Vascular disease is associated with facet joint osteoarthritis. Osteoarthritis Cartilage. 2010 Sep;18(9):1127-32. doi: 10.1016/j.joca.2010.06.012. Epub 2010 Jul 13. PMID 20633684